CLINICAL TRIAL: NCT03934476
Title: The Effects of Lowering Dietary Carbohydrates on Health, Exercise Performance and Wellbeing-related Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OU-PdF-GACR-LCHF diet; 18-08358S (Other Grant/Funding Number: GACR)
Record Dates: First submitted 2019-02-15; First posted 2019-05-01 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Diet Modification
Keywords: ketogenic diet; carbohydrates; chronic diseases; physical activity; fatigue; mood; wellbeing
MeSH Terms: conditions — Obesity; Chronic Disease; Motor Activity; Fatigue | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: The study subjects will be randomized into four study groups, one of which will be the control group.
Masking Description: No masking will be used in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ketogenic diet (Experimental): Ketogenic diet:
  * < 50 g carbohydrates - CHO/d (based on the 1-week pre-intervention habitual diet monitoring)
  * protein restriction ≤ 1.5 g/kg free-fat mass (FFM)/day.
  * fat type intake recommendation:
  * natural fats
  * trans-FA reduction
  Interventions: Behavioral: Ketogenic diet
- Exercise HIIT (High-Intensity Interval Training) (Experimental): Exercise intervention:
  - HIIT: 5 min warm-up - slow walking, 3 min interval of high-intensity walking (above VT2), 3 min interval of low-intensity walking (40 % VO2peak); 5 min cool-down - slow walking:
  Cycle 1
  * week 1-3 - 3 sessions/week, total time 31 min/session (4 intervals)
  * week 4 - regeneration: only 2 sessions with 2 intervals, keep total time 31 min/session, (+ GXT)
  Cycle 2
  * week 5-7 - 3 sessions/week, total time 43 min/session (6 intervals)
  * week 8 - regeneration: only 2 sessions with 4 intervals, total time 31 min/session, (+ GXT)
  Cycle 3
  * week 9-11 - 3 sessions/week, total time 55 min/session (8 intervals)
  * week 12 - regeneration: only 2 sessions with 6 intervals, total time 43min/session, (+GXT)
  Interventions: Behavioral: Exercise HIIT
- Ketogenic diet + Exercise HIIT (Experimental): Ketogenic diet:
  * < 50 g carbohydrates - CHO/d (based on the 1-week pre-intervention habitual diet monitoring)
  * protein restriction ≤ 1.5 g/kg free-fat mass (FFM)/day.
  * fat type intake recommendation:
  * natural fats
  * trans-FA reduction
  Exercise intervention:
  - HIIT: 5 min warm-up - slow walking, 3 min interval of high-intensity walking (above VT2), 3 min interval of low-intensity walking (40 % VO2peak); 5 min cool-down - slow walking:
  Cycle 1
  * week 1-3 - 3 sessions/week, total time 31 min/session (4 intervals)
  * week 4 - regeneration: only 2 sessions with 2 intervals, keep total time 31 min/session, (+ GXT)
  Cycle 2
  * week 5-7 - 3 sessions/week, total time 43 min/session (6 intervals)
  * week 8 - regeneration: only 2 sessions with 4 intervals, total time 31 min/session, (+ GXT)
  Cycle 3
  * week 9-11 - 3 sessions/week, total time 55 min/session (8 intervals)
  * week 12 - regeneration: only 2 sessions with 6 intervals, total time 43min/session, (+GXT)
  Interventions: Behavioral: Ketogenic diet; Behavioral: Exercise HIIT
- Control Group (No Intervention): The study subjects in this arm will undergo no dietary changes and no exercise intervention.

INTERVENTIONS:
Behavioral: Ketogenic diet — The study subjects randomized for this intervention will observe the ketogenic diet, as prescribed by the protocol.
  Arms: Ketogenic diet; Ketogenic diet + Exercise HIIT
Behavioral: Exercise HIIT — The study subjects randomized for this intervention will observe the HIIT exercise programme, as prescribed by the protocol.
  Arms: Exercise HIIT (High-Intensity Interval Training); Ketogenic diet + Exercise HIIT

SUMMARY:
The aim of the study is to investigate the long-term effects of the ketogenic diet and exercise (including interactions) on health markers, exercise performance and wellbeing outcomes in sedentary overweight individuals.

DETAILED DESCRIPTION:
Intentional nutritional ketosis induced by the low carbohydrate diet is an intensively discussed topic of many scientific as well as non-scientific discussions throughout the areas of healthy living, the sports sciences and often used now for the prevention and treatment of chronic diseases. It has been demonstrated that long-term low-carbohydrate diet is more effective for weight loss and cardiovascular and metabolic risk factor reduction than a low-fat diet. In light of conflicting theories of best practice surrounding a polarized topic that impacts human health and daily work performance, the primary aim of this research project is to examine how low-carbohydrate ketogenic diets affect health markers, exercise performance and wellbeing outcomes in sedentary overweight individuals. Each study subject will be randomized into one of the four arms of the study and will undergo a 12-week intervention, with the exception of the study subjects in the control group, who will undergo no intervention for the period of 12 weeks.

The project outcomes are of immense importance for the investigator's global human health, focus on a unique holistic perspective and have the potential to contribute towards much-needed adjustments in public health recommendations.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25.00 - 40.00 kg/m2
* non-smokers
* non-excessive alcohol intake (self-reported, ≥ to 2 drinks/day for men or ≥1 drink/day for women)
* willing to accept random assignment
* low active individuals over the last 1 year, i.e. no specific sports training or regular exercise (up to once a week) and self-reported physical activity < 150 min/week (IPAQ)
* no evidence of liver, renal, metabolic, and cardiopulmonary disease and dis-eases contraindicating physical activity, no cancer, no psychiatric illness
* Physical Activity Readiness Questionnaire (PAR-Q) pass
* body weight stable for the last 2 months and not actively on a weight loss plan
* prediabetes state allowed (impaired fasting glucose level, i.e. 5.6 - 6.9 mmol/l; HbA1c 5.7 - 6.4 %)

Exclusion Criteria:

* pregnancy, lactation
* any specific diet (e.g. vegetarian)
* use of hypoglycemic, lipid-lowering, antihypertensive, psychiatric medications or medications known to affect body weight or energy expenditure; any medication not noted allowed if the individual had been stable while taking such medication for at least 3 months prior to baseline data collection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the time to exhaustion | 12 weeks (baseline + every four weeks)
  All study subjects will undergo the Graded Exercise Test, with measuring of the time to exhaustion in minutes.
Change in cardiorespiratory variables - oxygen consumption | 12 weeks (baseline + every four weeks)
  All study subjects will undergo the Graded Exercise Test, with measuring of the oxygen consumption (L/min).
Change in cardiorespiratory variables - heart rate | 12 weeks (baseline + every four weeks)
  All study subjects will undergo the Graded Exercise Test, with measuring of the heart rate (beats per minute).

SECONDARY OUTCOMES:
Biochemical analysis - capillary blood | 12 weeks (2 times/week)
  All study subjects will undergo biochemical analysis of capillary blood - βHB and fasting glukose in mmol/L.
Biochemical analysis - venous blood | 12 weeks (2 times/week)
  All study subjects will undergo biochemical analysis of venous blood - oxidative stress, inflammation, total CHO, HDL, LDL, TG, FFA, GL, homocysteine, measured in mmol/L.
Biochemical analysis - venous blood | 12 weeks (2 times/week)
  All study subjects will undergo biochemical analysis of venous blood - HBA1c in mmol/mol.
Anthropometrics - body height | 12 weeks (baseline + every four weeks)
  All study subjects will undergo anthropometric assessment of the body height, measured in cm.
Anthropometrics - body weight | 12 weeks (baseline + every four weeks)
  All study subjects will undergo anthropometric assessment of the body weight, measured in kg.
Anthropometrics - waist circumference | 12 weeks (baseline + every four weeks)
  All study subjects will undergo anthropometric assessment of the waist circumference, measured in cm.
Anthropometrics - DXA | 12 weeks (baseline + outcome)
  All study subjects will undergo anthropometric assessment of DXA - total abdominal fat, measured in kg.
InBody (bioimpedance) | 12 weeks (baseline + every four weeks)
  All study subjects will undergo antrhropometric assessment of bioimpedance using the InBody device showing the percentage of water and fat in the organism, measured in % of total body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Lukáš Cipryan, Ass.Prof.,PhDr.,PhD, Principal Investigator — University of Ostrava
Locations (1):
- University of Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to share the individual participant data with other researchers.

REFERENCES:
- [Result] Cipryan L, Plews DJ, Ferretti A, Maffetone PB, Laursen PB. Effects of a 4-Week Very Low-Carbohydrate Diet on High-Intensity Interval Training Responses. J Sports Sci Med. 2018 May 14;17(2):259-268. eCollection 2018 Jun. PMID 29769827
- [Derived] Cipryan L, Kosek V, Garcia CJ, Dostal T, Bechynska K, Hajslova J, Hofmann P. A lipidomic and metabolomic signature of a very low-carbohydrate high-fat diet and high-intensity interval training: an additional analysis of a randomized controlled clinical trial. Metabolomics. 2023 Dec 23;20(1):10. doi: 10.1007/s11306-023-02071-1. PMID 38141101
- [Derived] Cipryan L, Litschmannova M, Maffetone PB, Plews DJ, Dostal T, Hofmann P, Laursen PB. Very Low-Carbohydrate High-Fat Diet Improves Risk Markers for Cardiometabolic Health More Than Exercise in Men and Women With Overfat Constitution: Secondary Analysis of a Randomized Controlled Clinical Trial. Front Nutr. 2022 May 23;9:867690. doi: 10.3389/fnut.2022.867690. eCollection 2022. PMID 35677551
- [Derived] Cipryan L, Dostal T, Litschmannova M, Hofmann P, Maffetone PB, Laursen PB. Effects of a Very Low-Carbohydrate High-Fat Diet and High-Intensity Interval Training on Visceral Fat Deposition and Cardiorespiratory Fitness in Overfat Individuals: A Randomized Controlled Clinical Trial. Front Nutr. 2021 Dec 21;8:785694. doi: 10.3389/fnut.2021.785694. eCollection 2021. PMID 34993222